CLINICAL TRIAL: NCT06618209
Title: Assessment of Oral Health Status of Children With Primary Ciliary Dyskinesia
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2023.305
Record Dates: First submitted 2024-09-04; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Primary Ciliary Dyskinesia; Caries,Dental; Quality of Life; Saliva Altered; Erosion, Dental Enamel
Keywords: primary ciliary dyskinesia; erosion, dental; oral health quality of life; dental caries
MeSH Terms: conditions — Ciliary Motility Disorders; Dental Caries; Tooth Erosion | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Children with primary ciliary dyskinesia group: It is a group of patients between the ages of 6 and 17 who have recently been diagnosed with primary ciliary dyskinesia
  Interventions: Diagnostic Test: physical and chemical methods; Diagnostic Test: biochemical methods; Diagnostic Test: Oral Findings; Diagnostic Test: Pediatric Oral Health Quality of Life
- healthy patient group: Healthy children aged between 6 and 17 years, with no systemic diseases and not taking any regular medications.
  Interventions: Diagnostic Test: physical and chemical methods; Diagnostic Test: biochemical methods; Diagnostic Test: Oral Findings; Diagnostic Test: Pediatric Oral Health Quality of Life
- Parents of children with Primary Ciliary Dyskinesia group: Parents of children aged 6-17 with Primary Ciliary Dyskinesia
  Interventions: Diagnostic Test: Pediatric Oral Health Quality of Life
- Parents of healthy children group: Parents of children aged 6-17 healthy children
  Interventions: Diagnostic Test: Pediatric Oral Health Quality of Life

INTERVENTIONS:
Diagnostic Test: physical and chemical methods — Salivary flow rate, pH
  Groups: Children with primary ciliary dyskinesia group; healthy patient group
Diagnostic Test: biochemical methods — Total oxidant and antioxidant capacities, Lactoperoxidase, Oxidative Stress Index, Glutathione, Superoxide Dismutase
  Groups: Children with primary ciliary dyskinesia group; healthy patient group
Diagnostic Test: Oral Findings — DMFT/dft Index: Measures decayed, missing, and filled teeth. ICDAS II: International Caries Detection and Assessment System, used for detecting and assessing dental caries. DDE Index: Developmental Defects of Enamel index.GI (Gingival Index): Assesses the severity of gingivitis based on inflammation.PI (Plaque Index): Assesses the severity of plaque based on inflammation. basic erosive wear examination: measures dental erosion
  Groups: Children with primary ciliary dyskinesia group; healthy patient group
Diagnostic Test: Pediatric Oral Health Quality of Life — The Pediatric Oral Health Quality of Life (POQL) Scale is a tool used to assess the impact of oral health conditions on the overall quality of life in children.

SUMMARY:
The aim of this study is to compare the oral health findings, salivary parameters and pediatric oral health related quality of life of children with Primary Ciliary Dyskinesia (PCD) with healthy children

DETAILED DESCRIPTION:
Primary Ciliary Dyskinesia (PCD) is a rare genetic disorder that affects the function of cilia, which are tiny hair-like structures responsible for moving mucus and other substances in the respiratory tract and other parts of the body. Dysfunctional cilia lead to impaired mucociliary clearance, resulting in chronic respiratory infections, sinusitis, and bronchiectasis. PCD can also cause situs inversus, where internal organs are mirrored from their normal positions, and other complications like chronic otitis media and fertility issues. Early diagnosis and management are crucial to prevent progressive lung damage and improve the quality of life in affected individuals.

This study aims to compare the oral and dental health of children diagnosed with Primary Ciliary Dyskinesia (PCD) to that of healthy controls. The study includes assessments of dental caries (using DMFT, dmft, and ICDAS II indices), salivary parameters (flow rate, pH, buffering capacity, oxidant-antioxidant levels, tissue factor activity), enamel defects (using the Modified Developmental Defects of Enamel Index), and oral hygiene (gingival and plaque indices). The Pediatric Oral Health-Related Quality of Life (POQL) scale will be used to evaluate the impact of oral health on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Not having any systemic disease.
* Not being on any regular medication.

Exclusion Criteria:

* Having any systemic disease.
* Being on any regular medication.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Being followed up for a diagnosis of primary ciliary dyskinesia
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life (QoL) | baseline
  The Pediatric Oral Health Quality of Life (POQL) Scale is used to measure how oral heThe Pediatric Oral Health Quality of Life (POQL) Scale measures the impact of oral health on a child's quality of life. Scores range from 0 to 100, with higher scores indicating a worse outcome, reflecting a greater negative impact of oral health on daily life and well-being.alth impacts a child's daily activities, well-being, and overall quality of life.
Oral Health Status: DMFT/dft Index | baseline
  DMFT/dft Index: Reported as numerical values representing the number of decayed (D), missing (M), and filled (F) teeth in the permanent (DMFT) and primary (dft) dentition. These values will reflect the overall dental health of participants by quantifying the extent of caries and treatment.
Oral Health Status: Gingival Index (GI) | baseline
  Gingival Index (GI): Reported as numerical values indicating the severity of gingival inflammation. GI scores range from 0 (healthy) to 3 (severe inflammation), giving insight into the participants' gum health.
Oral Health Status: Developmental Defect of Enamel (DDE) Index | baseline
  Developmental Defect of Enamel (DDE) Index: Presented as the percentage of participants with observed enamel defects. This percentage helps quantify how many children experience developmental issues affecting enamel quality.
Oral Health Status: Basic Erosive Wear Examination (BEWE) | baseline
  Basic Erosive Wear Examination (BEWE): Reported as the percentage of participants showing signs of erosive tooth wear. The BEWE score categorizes wear and provides a general picture of tooth surface loss due to erosion.
Oral Health Status: International Caries Detection and Assessment System (ICDAS-II) | baseline
  International Caries Detection and Assessment System (ICDAS-II): Expressed as the percentage of participants with caries at various stages, from early demineralization to advanced decay. This system provides a nuanced view of the caries progression within the population.
Salivary Analysis: Glutathione (GSH) and Lipid Peroxidation (LPO) | baseline
  Glutathione (GSH): Reported in µmol/L, measuring the concentration of this antioxidant. Lipid Peroxidation (LPO): Reported in µmol/L as malondialdehyde equivalents, indicating lipid peroxidation.
Salivary Analysis: Total Antioxidant Status (TAS) | baseline
  Total Antioxidant Status (TAS): Measured in µmol Trolox/L, indicating the saliva's antioxidant capacity.
Salivary Analysis: Total Oxidant Status (TOS) | baseline
  Total Oxidant Status (TOS): Expressed in µmol H₂O₂/L, reflecting oxidative stress in saliva.
Salivary Analysis: Salivary Flow Rate | baseline
  Salivary Flow Rate: Measured in mL/min, representing the volume of saliva produced.
Salivary Analysis: Superoxide Dismutase (SOD) | baseline
  Superoxide Dismutase (SOD): Reported in U/mg protein, showing enzyme activity in neutralizing superoxide radicals.
Salivary Analysis: Oxidative Stress Index (OSI) | baseline
  Oxidative Stress Index (OSI): Calculated as the ratio of TOS to TAS, representing oxidative stress.
Oral Health Status: Plaque Index (PI) | baseline
  Plaque Index (PI): Also reported as numerical values, representing the amount of plaque accumulation on the teeth. Like the GI, PI helps assess oral hygiene levels.

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Karadag, Study Chair — Marmara University Faculty of Medicine; Ela Erdem Eralp, Study Chair — Marmara University Faculty of Medicine; Yasemin Gokdemir, Study Chair — Marmara University Faculty of Medicine
Locations (1):
- Marmara University Faculty of Dentistry, Istanbul, Maltepe, Turkey (Türkiye)

REFERENCES:
- [Derived] Oztuna EK, Peker S, Eralp EE, Gokdemir Y, Karadag B. Oral Health Status and Oral Health-Related Quality of Life in Children With Primary Ciliary Dyskinesia. Pediatr Pulmonol. 2025 Nov;60(11):e71370. doi: 10.1002/ppul.71370. PMID 41221835